CLINICAL TRIAL: NCT06077487
Title: Pilot Study of Ketamine-assisted Talk Therapy for Demoralization in Advanced GI Cancer
Brief Title: Ketamine-assisted Therapy for Advanced GI Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Brian Anderson, MD (Other)
Responsible Party: Sponsor-Investigator, Brian Anderson, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 238011; NCI-2023-07386 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Pain, Acute; Gastrointestinal Cancers; Demoralization
Keywords: Medication assisted therapy; ketamine
MeSH Terms: conditions — Acute Pain; Gastrointestinal Neoplasms | interventions — Ketamine; Psychotherapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is double-blinded, meaning neither the study participants nor the study investigators will know which ketamine administration each participant is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Blinded Group A (K-MaP) (Experimental): Participants will receive 0.5mg/kg of Ketamine orally with an equivalent quantity of placebo via an intramuscular injection on Day 0/Visit 4 and receive Meaning and Purpose (MaP) therapy 4 times, twice before (between days -13 and -1) ketamine administration, and twice afterward on days 3 (+/- 2 days) and 11 (+/- 3 days). The duration of treatment for ketamine plus MaP (K-MaP) therapy is approximately up to 28 days. Participants will be followed up to 35 days (+/-2 days) after ketamine administration.
  Interventions: Drug: Ketamine; Behavioral: Meaning and Purpose therapy; Other: Placebo; Other: Questionnaires
- Blinded Group B (K-Map) (Experimental): Participants will receive 0.5mg/kg of Ketamine IM with a placebo oral solution on Day 0/Visit 4 and receive Meaning and Purpose (MaP) therapy 4 times, twice before (between days -13 and -1) ketamine administration, and twice afterward on days 3 (+/- 2 days) and 11 (+/- 3 days). The duration of treatment for ketamine plus MaP (K-MaP) therapy is approximately up to 28 days. Participants will be followed up to 35 days (+/-2 days) after ketamine administration.
  Interventions: Drug: Ketamine Injectable Product; Behavioral: Meaning and Purpose therapy; Other: Placebo; Other: Questionnaires

INTERVENTIONS:
Drug: Ketamine — Given orally (PO)
  Other Names: Ketalar; Ketalar Hydrocholoride
  Arms: Blinded Group A (K-MaP)
Drug: Ketamine Injectable Product — Given intramuscularly (IM)
  Other Names: Ketalar; Ketalar Hydrocholoride
  Arms: Blinded Group B (K-Map)
Behavioral: Meaning and Purpose therapy — In-person sessions
  Other Names: MaP; MaP therapy; Psychotherapy
Other: Placebo — Given PO or IM
Other: Questionnaires — Questionnaires will be given over the course of the study

SUMMARY:
This clinical trial evaluates whether it is possible to use a single dose of ketamine in combination with talk therapy to treat moderate to severe demoralization in patients with stage 3 or 4 gastrointestinal (GI) cancers who take opioids for cancer-related pain. Advanced stage gastrointestinal (GI) cancer patients often suffer from high rates of psychosocial distress and pain. Symptoms of anxiety are highly prevalent among gastrointestinal (GI) cancers patients. While opioid analgesia (pain reliever) succeeds in managing some symptoms, chronic opioid therapy is associated with significant adverse effects, underscoring a need to identify alternative interventions in the treatment of cancer associated pain. GI cancer patients frequently suffer from existential distress, and demoralization is a form of existential distress that is common among people with serious medical illnesses. Demoralization is characterized by poor coping with stressful events, and a loss of meaning and purpose in life. Talk therapy is a form of psychological treatment during which patients discuss problems, thoughts, and feelings. Ketamine has demonstrated efficacy for the treatment of depression, suicidality, and pain in non-cancer patients. This study may help researchers learn whether ketamine and talk therapy combined may improve psychosocial distress and pain, as well as decreases opioid analgesic use in patients with advanced GI cancer who take opioids for cancer-related pain.

DETAILED DESCRIPTION:
PRIMARY OUTCOMES:

I. To assess the feasibility of Meaning and Purpose therapy combined with oral ketamine (K-MaP) in demoralized participants.

SECONDARY OUTCOMES:

I. To characterize the preliminary safety and tolerability of K-MaP in demoralized participants with stage 3 or 4 gastrointestinal (GI) cancers.

II. To assess the magnitude and durability of improvement from randomization in psychosocial distress.

III. To assess the magnitude and durability of improvement from randomization in pain.

IV. To assess the magnitude of change from randomization in opioid analgesic use.

V. To assess the magnitude and durability of change from randomization in interoceptive awareness

EXPLORATORY OBJECTIVES:

I. To assess how the participant's subjective experiences with ketamine may be related to clinical outcomes.

II. To assess how participants' stage of cancer may be related to clinical outcomes.

III. To assess how the participants' changes in measures of cardiac interoception following receipt of ketamine may be related to subjective experiences with ketamine and clinical outcomes.

OUTLINE:

Adult participants with advanced stage GI cancers receiving care at the Helen Diller Family Comprehensive Cancer Center (HDFCCC) will be randomized in a 1:1 ratio to one of two double-blinded conditions consisting of a single drug treatment and several therapy sessions. Participants will be followed up to 35 days (+/-2 days) after ketamine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a diagnosis of a stage 3 or 4 primary GI (i.e., pancreatic, colorectal, hepatocellular, biliary, and gastro-esophageal) cancer.
2. Must be willing to sign the informed consent form (ICF) and follow the study procedures as outlined in the ICF for the duration of the study.
3. Must be 18 years or older.
4. Must speak English and/or Spanish
5. Must have a Palliative Performance Score (PPS) v. 2.0 greater than or equal to 40%.
6. Must be able to swallow liquid oral medication.
7. Clinically significant moderate to severe demoralization as assessed by the Demoralization Scale-II (DS-II).
8. Must discontinue the following medications and refrain from taking following medications for the duration of study participation (participants who require these medications will be taken off study):

   1. Lamotrigine
   2. Clozapine
   3. as-needed (PRN) anxiolytics. Note: Benzodiazepine use may be allowed if used in a regular, scheduled way. Consultation with the Principal Investigator is recommended.
   4. Dopamine agonists
   5. Lithium
9. Female-born participants of child-bearing potential with male-born partners must use highly effective contraception for at least 1 month prior to ketamine administration (on day 0) and agree to use such a method for an additional 2 months after ketamine administration.
10. Male-born participants with female-born partners of child-bearing potential must use highly effective contraception for at least 1 month prior to ketamine administration and agree to use such a method for an additional 2 months after ketamine administration. Note: Highly effective contraception include:

    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Non-oral hormonal methods, including injected, intravaginal, implanted, transdermal
    * Oral hormones plus a barrier contraception (condom, diaphragm, or spermicide)
    * Double barrier method (at least two of the following: condom, diaphragm, and spermicide)
    * Vasectomy
    * Abstinence from penile-vaginal intercourse* *The reliability of abstinence should be evaluated carefully with the participant in relation to their general lifestyle. An additional acceptable birth control method should be discussed with the participant in case participants decide to engage in penile-vaginal intercourse during the course of the study.
11. Must agree to the following life-style considerations:

    1. Continue receiving psychotherapy or other behavioral interventions for mental health as usual. Current interventions should not be stopped and new interventions should not be started during the study period once participants are enrolled in the study.
    2. Consume no more than a modest quantity (e.g., 1 cup) of caffeine or xanthine-containing products (e.g., coffee or tea) the morning of receiving ketamine (on Day 0/Visit 4).
    3. Abstain from alcohol for 24 hours before receiving ketamine.
    4. Abstain from using any nicotine-containing products (including nicotine patches) for 3 hours before receiving ketamine.
    5. If cannabis products are used regularly, participants will be asked to continue using regular amount but will be asked not to use cannabis within 24 hours prior to receiving ketamine.
    6. If prescribed a regular dose of benzodiazepines, participants will be asked not to take medication the morning of the ketamine administration visit.
    7. If taking any psychostimulants (e.g., methylphenidate), participants will be asked not to take psychostimulant drugs (other than caffeine) the morning of the ketamine administration visit.
    8. Will be advised to maintain their usual opioid regimen.

Note: Input will be obtained from the participant's regular clinical providers on appropriate pain management for the participant during the study, particularly in the case of analgesics associated with adverse reactions of concern with ketamine (e.g., tramadol and any opioid may increase risk of respiratory depression from ketamine).

Exclusion Criteria:

1. Has a known allergic or severe reactions to the non-psychoactive components of liquid ketamine.
2. Has received treatment with another investigational drug or intervention within 1 month of signing Informed Consent Form (ICF).
3. Is deemed by clinical judgment of the study investigators to be unsafe for undergoing the intervention.
4. Recent use of ketamine for non-anesthesia purposes.
5. Frequent use of ketamine over lifetime.
6. Has a history of intra-cerebral hemorrhage.
7. Has cognitive impairment sufficient to impede the ability to complete study tasks.
8. Has had delirium/encephalopathy within 3 months of signing ICF.
9. Has a history of intracranial hemorrhage.
10. Has had a stroke (embolic) within 12 months of signing ICF.
11. Has had a seizure within 6 months of signing ICF.
12. Currently has an intracranial mass (e.g., primary tumor or brain metastasis).
13. Has an advanced stage of a neurologic disease that puts participants at elevated risk for psychosis (e.g., Parkinson or Huntington disease).
14. Has a history of a primary psychotic disorder or primary bipolar disorder I or II (determined by Quick Structured Clinical Interview for Diagnostic and Statistical Manual version 5 Disorders (QuickSCID-5)).
15. Has a history of dissociative disorder.
16. Recent active suicidal ideation. Note: This does not include requesting medical aid in dying.
17. Is currently receiving electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS) or similar somatic therapies.
18. Has baseline hypertension (≥150 SBP or ≥90 DBP), after repeated measurements. Note: Participants with hypertension that has been controlled by medication down to <150 Systolic blood pressure (SBP) and <90 diastolic blood pressure (DBP) will be allowed participate.
19. Has a history of aneurysmal vascular disease or dissection (including thoracic and abdominal aorta, intracranial and peripheral arterial vessels) or arteriovenous malformation.
20. Has had cardiac arrest within 12 months of signing ICF.
21. Has had a myocardial infarction within 12 months of signing ICF.
22. Has QT Corrected for Heart Rate using Fridericia's Formula (QTcf) >480msec on 12-lead EKG. Note: Participants may qualify for the study if corrected QT Interval (QTc) 480-500 msec on one EKG, but then <=480 msec on repeat EKG taken >1 day later. If QT-prolonging medications are started or increased in dose after enrollment and prior to ketamine administration, a repeat EKG must be done >12-hours after this change in order to assure continued safe enrollment in the trial.
23. Has clinically significant arrhythmia defined as

    1. Ventricular fibrillation or ventricular tachycardia within 1 year of signing ICF
    2. Bradycardia, severe, within 1 year of signing ICF Note: Participants with pacemakers will be considered to be eligible at the discretion of the Principal Investigator.
    3. Atrial fibrillation, without rate or rhythm control
    4. Supraventricular tachycardia (SVT), without standard treatment
    5. Other clinically significant arrhythmias (e.g., Wolf Parkinson White)
24. Has symptomatic congestive heart failure (NYHA Class II-IV)
25. Has severe obstructive intracardiac abnormalities (e.g., aortic stenosis)
26. Has any current condition where physical activity is associated with palpitations, anginal pain or syncope.
27. Is unable to protect their own airway due to dysphagia, difficulty swallowing or a neurologic disease resulting in a risk of aspiration.
28. Has a history of flash pulmonary edema within 12 months of signing ICF.
29. Has a diagnosis of moderate or severe pulmonary hypertension.
30. Needs supplemental oxygen (intermittent or continuous).
31. Has current intractable nausea/vomiting/diarrhea.
32. Meets the following laboratory parameters:

    1. Asymptomatic alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >=5x upper limit of normal (ULN).
    2. Symptomatic ALT or AST >= 2x ULN.
    3. Total bilirubin > 2x ULN (Gilbert syndrome is allowed)
    4. Alkaline phosphatase >5x ULN
    5. International Normalized Ratio (INR) > 2.5 for patients with any history of cirrhosis or gastrointestinal bleeding within 6 months of signing ICF.
    6. Renal insufficiency (i.e., estimated glomerular filtration rate (eGFR) < 30 milliliter/minute (mL/min) /1.73 m^2 (using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation), Creatinine Clearance (CrCl) < 30 mL/min (using the Cockcroft-Gault Equation), or current dialysis)).
33. Is currently pregnant or breastfeeding.
34. Has insulin-dependent diabetes with diabetes-related hospitalization within 6 months of signing ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian T Anderson, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were pre-screened via phone prior to signing consent to determine if eligible for a visit to sign the informed consent in person. Once consent was signed, those participants were assigned to 1 of 2 blinded conditions. Only 1 person who was eligible signed consent and was assigned to a blinded arm of the study.
Period: Overall Study
Arm/Group | Blinded Group A (K-MaP) | Blinded Group B (K-Map)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only 1 participant was enrolled on this protocol. No participants meet the criteria to be considered evaluable for this protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Group A (K-MaP) | Blinded Group B (K-Map) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Count of Participants; unit: Participants]
  70-79 years old |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion Eligible Versus Screened Participants.
Description: The rate of recruitment is defined as the proportion of eligible participants who participate compared to the number of total participants who were screened or signed consent but did not meet eligibility criteria will be reported.
Time Frame: Up to 28 days
Measure: Number; unit: proportion of potential participants
Groups:
- Screened Participants: Potential participants will be screened by phone to determine if they will be eligible for a visit to sign informed consent for blinded portion of the study.
Arm/Group | Screened Participants
Number analyzed (Participants) | 5
proportion of potential participants | .60

2. Primary Outcome: Proportion of Participants Who Complete Therapy
Description: Proportion of enrolled participants completing K-MaP intervention and all Demoralization Scale II (DS-II) assessments will be reported.
Time Frame: Up to 49 days
Measure: Number; unit: participants
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 1
participants | 0

3. Primary Outcome: Frequency of Participant Responses to Intervention Acceptability
Description: The participants will provide qualitative feedback on the acceptability of the intervention via a 20-minute interview with the study team upon study termination. Frequency of responses will be categorized and reported by arm.
Time Frame: 1 day
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants Reporting Treatment-emergent Adverse Events
Description: The percentage of participants in each arm reporting treatment-related adverse events will be reported. Pre-determined criteria for assessment of tolerability to K-MaP include zero treatment-related serious adverse events, and all other adverse events will be assessed using Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to 49 days
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 1
percentage of participants | 100

5. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Blood Pressure
Description: At time of ketamine administration, participants blood pressure will be monitored for any clinically significant changes. The percentage of participants with a clinically significant change in blood pressure from pre-medication administration to end of study visit will be reported.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 1
percentage of participants | 100

6. Secondary Outcome: Percentage of Participants With Clinically Significant Changes in Heart Rate
Description: At time of ketamine administration, participants heart rate will be monitored for any clinically significant changes. The percentage of participants with a clinically significant change in heart rate from pre-medication administration to end of study visit will be reported.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 1
percentage of participants | 0

7. Secondary Outcome: Mean Scores on the Challenging Experience Questionnaire (CEQ) Over Time
Description: The CEQ is a 26-item, self-reported measure of challenging experiences with psychedelics. The CEQ assesses seven factors: grief (5 items), fear (6 items), subjective experience of death (2 items), insanity (3 items), isolation (3 items), physical distress (5 items), and paranoia (2 items). Each of the 26 items is scored on a 5-point Likert scale (0 = "None; not at all" to 5 = "Extreme [more than ever before in my life]"). Participants are asked to rate each item based on the degree to which each item was experienced. A higher total CEQ score indicates greater psychologically adverse reactions to psilocybin.
Time Frame: 1 day
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

8. Secondary Outcome: Mean Clinician-rated Scores on the Global Clinical Impression of Severity (CGI-S) Over Time
Description: The CGI is a 3-item clinician-administered measure developed by the National Institute of Mental Health to assess clinical change in participants in psychopharmacology trials. This study will be using the Global Impression of Severity item ("Considering your total clinical experience with participants with demoralization, how would you rate this participant's level of demoralization at this time?"), on the scale from "1 = Normal, not at all demoralized" to "7 = Among the most extremely demoralized participants" to assess change in demoralization.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Clinician-rated Scores on the Demoralization Interview (DI) Over Time
Description: The DI is a clinician-rated measure of demoralization which consists of 14-items designed from items of the Demoralization Scale II. The items measure events that occurred over the past 2 weeks, which are scored on a 3-point scale ranging from 0 to 2. Scores are calculated by adding each item score, for a total score range of 0 to 28. Higher scores indicate a greater degree of demoralization.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

10. Secondary Outcome: Mean Clinician-rated Scores on the GRID-Hamilton Depression Rating Scale (GRID-HAMD) Over Time
Description: The 6-item Hamilton Depression Rating Scale (HAMD-6) is a validated, brief, clinician-rated measure of the core symptoms of major depression. With permission from authors (the International Society for Central Nervous System Drug Development (ISCDD)) a modified, 6-items version of the HAMD-6 in the GRID-HAMD format to will be used by clinicians to create a brief, responsive and reliable measure of core depression symptoms of participants. Responses on the items will range from 0=absent; 1=mild; 2=moderate; 3=severe; 4=incapacitating and scores will be summed to create a total score. The higher the total score the more severe the depression symptoms of the participant.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

11. Secondary Outcome: Proportion of Participants With Reported Demoralization Based on the Diagnostic Criteria in Psychosomatic Research (DCPR) Demoralization Scale.
Description: The DCPR is a structured, clinician-administered, interview regarding various psychosomatic conditions and will be administered to participants over the course of the study. Clinicians will record the rates of demoralization as present or not per participant
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

12. Secondary Outcome: Mean Scores on the Demoralization Scale II (DS-II) Over Time
Description: The DS-II is a measure of demoralization which consists of 16-items designed from items of the Demoralization Scale II. The items measure events that occurred over the past 2 weeks, which are scored on a 3-point scale ranging from 0 to 2. Scores are calculated by adding each item score, for a total score range of 0 to 32. Higher scores indicate a greater degree of demoralization.
Time Frame: Up to 49 days
Population: Data not collected
Groups:
- Group B (K-Map): Participants will receive 0.5mg/kg of Ketamine IM with a placebo oral solution on Day 0/Visit 4 and receive Meaning and Purpose (MaP) therapy 4 times, twice before (between days -13 and -1) ketamine administration, and twice afterward on days 3 (+/- 2 days) and 11 (+/- 3 days). The duration of treatment for ketamine plus MaP (K-MaP) therapy is approximately up to 28 days. Participants will be followed up to 35 days (+/-2 days) after ketamine administration.
Arm/Group | Group B (K-Map)
Number analyzed (Participants) | 0

13. Secondary Outcome: Mean Scores on the Patient Health Questionnaire 9 (PHQ-9) Over Time
Description: The Patient Health Questionnaire-9 (PHQ-9) is used to measure depression symptoms. The total Patient Health Questionnaire-9 (PHQ-9) score is calculated by combining the responses of the participant on questions addressing how bothered the participant has been by various problems over the past 2 weeks. Each of the 9 items is scored on a scale of 0 ("Not bothered at all") to 4 ("Nearly every day"). A total score of 5-9='Mild Depression Symptoms", 10-14="Minor Depression, Major Depression (mild), or Dysthymia", 15-19="Major Depression, moderately severe", and >20="Major Depression".
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

14. Secondary Outcome: Mean Scores on the Generalized Anxiety Disorder 7 (GAD-7) Over Time
Description: The GAD-7 is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder. The GAD-7 score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of "not at all," "several days," "more than half the days," and "nearly every day," respectively, and then adding together the scores for the seven questions. Scores of 5, 10, and 15 represent cut-points for mild, moderate, and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

15. Secondary Outcome: Mean Scores on the Functional Assessment of Chronic Illness Therapy Palliative Care, 14 Item Version (FACIT-Pal-14) (FACIT-Pal-14) Over Time
Description: The FACIT-Pal-14 is a 14-item, self-report measure of quality of life in palliative care participants. The measure has a 7-day recall period with responses to items which fall on a 5-point Likert scale, with scores ranging from 0 = "Not at all" to 4 = "Very much". Scores are summed to create a total score of 0 to 56, with higher scores indicating a greater quality of life.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

16. Secondary Outcome: Mean Scores on the Brief-Pain Inventory Short Form (BPI-SF) Over Time
Description: The BPI-SF is a 9-item questionnaire used to assess the severity of pain and the impact of pain on activities of daily living over a recall period of 24 hours. Pain severity is assessed across four sub-scales; 'worst pain', 'least pain', 'average pain' and 'current pain'. A pain score for each subscale is presented separately. Scales are rated on a scale of 0 to 10 (0 = no pain; 10 = pain as bad as one can imagine). A composite score for pain severity is calculated as the mean of the four severity items. Question 9 comprises a 7-item interference scale. Questions assess the level to which pain interferes with general activity, walking, work, mood, enjoyment of life, relations with others and sleep on a scale of 0 to 10 (0 = does not interfere; 10 = completely interferes). Mean interference score will be calculated as an average of the seven subparts of question 9 where at least four of the seven items are completed.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

17. Secondary Outcome: Proportion of Participants Reporting Any Use of Prescribed Opioids
Description: The proportion of participants with any reported prescribed opioid use at any of the study visits will be reported.
Time Frame: Up to 49 days
Measure: Number; unit: proportion of participants
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 1
proportion of participants | 1.00

18. Secondary Outcome: Mean Scores on the Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2)
Description: The MAIA-2 is a validated a widely used questionnaire to measure interoceptive awareness. This measure consists of 37-items using a 6-point Likert scale (0 = "Never" to 5 = "Always"). The MAIA-2 has demonstrated good internal consistency and reliability for the evaluation of clinical mind-body interventions, with higher scores indicating increased awareness.
Time Frame: Up to 49 days
Population: Data not collected
Arm/Group | Blinded Group B (K-Map)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Only 1 participant was enrolled in the study. Serious Adverse Events were unrelated to intervention, and only 2 adverse events (feeling 'energized' and paresthesia) were attributable to the study intervention.
Arm/Group | Blinded Group A (K-MaP) | Blinded Group B (K-Map)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Group A (K-MaP) (N=0) | Blinded Group B (K-Map) (N=1)
Transient Ischemic Attack (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Group A (K-MaP) (N=0) | Blinded Group B (K-Map) (N=1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) — Metallic taste in mouth
Hypertension (Vascular disorders) | 0 (0) | 1 (1) — Elevated blood pressure
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders, Other (Nervous system disorders) | 0 (0) | 1 (1) — Energized

LIMITATIONS AND CAVEATS:
The study was terminated after one accrual due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT06077487/Prot_SAP_000.pdf